CLINICAL TRIAL: NCT00002610
Title: National Wilms Tumor Study-5 -- Treatment of Relapsed Patients, A National Wilms Tumor Study Group Phase III Study
Brief Title: Chemotherapy With or Without Surgery, Radiation Therapy, or Stem Cell Transplantation in Treating Young Patients With Kidney Tumors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Purpose: Treatment
Other Study IDs: 9444; COG-Q9402 (Other: Children's Oncology Group); NWTS-Q9402 (Other: NWTS); CCG-4942 (Other: Children's Cancer Group); POG-9444 (Other: Pediatric Oncology Group); INT-0152; NWTS-5/R (Other: NWTS); CDR0000063900 (Other: NCI)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Kidney Cancer
Keywords: recurrent Wilms tumor and other childhood kidney tumors; clear cell sarcoma of the kidney; rhabdoid tumor of the kidney
MeSH Terms: conditions — Kidney Neoplasms; Wilms Tumor | interventions — Dactinomycin; Filgrastim; Granulocyte Colony-Stimulating Factor; Carboplatin; Cyclophosphamide; Doxorubicin; Etoposide; Vincristine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- STRATUM A (Experimental): Treatment of children in Stratum A will be determined by the site of relapse and the presence of microscopic or gross residual disease after attempted surgical excision of the relapse.
  Interventions: Biological: dactinomycin; Drug: doxorubicin hydrochloride; Drug: vincristine sulfate; Procedure: conventional surgery; Radiation: radiation therapy
- Stratum B (Experimental): All children who received combination chemotherapy with Regimen EE - 4A as their initial therapy for Wilms tumor will receive Regimen I and radiation therapy to the site of recurrence. All patients will receive prophylactic trimethoprim /sulfamethoxazole
  Interventions: Biological: filgrastim; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: vincristine sulfate; Procedure: conventional surgery; Radiation: radiation therapy
- STRATUM C (Experimental): All children who received combination chemotherapy with Regimen DD - 4A as their initial therapy for Wilms tumor will be treated with the following chemotherapy. All patients will receive prophylactic trimethoprim/sulfamethoxazole
  Interventions: Biological: filgrastim; Drug: carboplatin; Drug: cyclophosphamide; Drug: etoposide; Procedure: conventional surgery; Radiation: radiation therapy
- STRATUM D (Experimental): Six week cycles of chemotherapy will be given to all patients who do not have progressive disease at the time of each week 0 re-evaluation.
  Interventions: Drug: carboplatin; Drug: etoposide

INTERVENTIONS:
Biological: dactinomycin
  Other Names: Actinomycin-D; Cosmegen; NSC #3053
  Arms: STRATUM A
Biological: filgrastim
  Other Names: Granulocyte-colony stimulating factor; r-MetHuG-CSF; GCSF; Neupogen; NSC #614629
  Arms: STRATUM C; Stratum B
Drug: carboplatin
  Other Names: CBDCA; NSC #241240
  Arms: STRATUM C; STRATUM D
Drug: cyclophosphamide
  Other Names: CTX; Cytoxan; NSC #2626-71
  Arms: STRATUM C; Stratum B
Drug: doxorubicin hydrochloride
  Other Names: Adriamycin; NSC #123127
  Arms: STRATUM A; Stratum B
Drug: etoposide
  Other Names: VP-16; VePesid; NSC #141540
  Arms: STRATUM C; STRATUM D; Stratum B
Drug: vincristine sulfate — IV
  Other Names: VCR
  Arms: STRATUM A; Stratum B
Procedure: conventional surgery
  Arms: STRATUM A; STRATUM C; Stratum B
Radiation: radiation therapy
  Arms: STRATUM A; STRATUM C; Stratum B

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells. It is not yet known which therapy regimen is most effective for treating patients with kidney tumors.

PURPOSE: Phase III trial to compare the effectiveness of chemotherapy with or without radiation therapy, surgery, and/or peripheral stem cell or bone marrow transplantation in treating young patients with kidney tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the 2-year second-event-free survival after vincristine (VCR) and dactinomycin (DACT) with or without doxorubicin (DOX), depending on the site of relapse and presence of microscopic residual disease, in children with relapsed Wilm's tumor previously treated with nephrectomy alone as initial therapy.
* Determine whether the 2-year second-event-free survival after intensive doxorubicin, etoposide (VP-16), cyclophosphamide (CTX), and carboplatin (CBDCA) plus radiotherapy to residual disease is at least 40% higher in patients with relapsed Wilm's tumor previously treated with Regimen EE-4A as initial therapy and without loss of heterozygosity for chromosomes 16q and 1p and increased DNA content in tumor cells than for similarly treated patients with loss of heterozygosity for chromosome 16q or 1p or increased DNA content in tumor cells.
* Determine whether the 4-year post-relapse survival after intensive VP-16, CTX, and CBDCA is at least 40% higher in patients with relapsed Wilm's tumor previously treated with Regimen DD-4A as initial therapy and without loss of heterozygosity for chromosomes 16q and 1p and increased DNA content in tumor cells than for similarly treated patients with loss of heterozygosity for chromosome 16q or 1p or increased DNA content in tumor cells.
* Determine whether the rates of complete and partial response exceed 20% in patients with relapsed clear cell sarcoma of the kidney or diffuse anaplastic Wilms' tumor treated with CBDCA combined with VP-16.

OUTLINE: This is a multicenter study.

Patients are assigned to a treatment group based on initial therapy and histology. Patients under age 2 at diagnosis who were previously treated with nephrectomy as initial therapy for stage I favorable histology Wilms' tumor weighing less than 550 grams are assigned to group A. Patients who received Regimen EE-4A as initial therapy for Wilms' tumor are assigned to group B. Patients who received Regimen DD-4A as initial therapy for Wilms' tumor are assigned to group C. Patients with clear cell sarcoma of the kidney or diffuse anaplastic Wilms' tumor are assigned to group D.

Group A

* Treatment is determined by site of relapse and the presence of microscopic or gross residual disease after attempted resection of relapsed disease. Children with suspected intra-abdominal recurrence undergo exploratory surgery to determine the site of recurrence and to obtain tissue for microscopic examination. Patients with stage I disease after recurrence are treated with regimen EE-4A. Patients with stage II or III disease are treated with regimen DD-4A.

  * Regimen EE-4A: Patients receive dactinomycin (DACT) IV on weeks 0, 3, 6, 9, 12, 15, and 18 and vincristine (VCR) IV on weeks 1-10, 12, 15, and 18 in the absence of disease progression.
  * Regimen DD-4A: Patients receive DACT IV on weeks 0, 6, 12, 18, and 24; VCR IV weekly on weeks 1-10, 12, 15, 18, 21, and 24; doxorubicin (DOX) IV on weeks 3, 9, 15, and 21; and abdominal radiotherapy in the absence of disease progression.

Group B

* Patients undergo resection. After resection, patients receive regimen I comprising DOX IV on weeks 0, 6, 12, 18, and 24; VCR IV on weeks 1, 2, 4, 5-8, 10-13, 18, and 24; cyclophosphamide (CTX) IV over 1 hour on days 1-3 of weeks 6, 12, 18, and 24 and on days 1-5 of weeks 3, 9, 15, and 21; and etoposide (VP-16) IV over 1 hour (after CTX infusion) on days 1-5 of weeks 3, 9, 15, and 21 in the absence of disease progression. Filgrastim (G-CSF) is administered subcutaneously (SC) beginning 24 hours after completion of chemotherapy and continuing until blood counts recover. Patients undergo radiotherapy to site of recurrence beginning within 1 week after initiation of chemotherapy.

Group C

* Induction: Patients receive CTX IV over 1 hour on days 1-5 of weeks 0 and 3; VP-16 IV over 1 hour (after CTX infusion) on days 1-5 of weeks of 0 and 3 and on days 1-3 of weeks 6 and 9; and carboplatin (CBDCA) IV over 6 hours on days 1 and 2 of weeks 6 and 9 in the absence of disease progression. G-CSF is administered SC beginning 24 hours after completion of CTX/VP-16 or CBDCA/VP-16 and continuing until blood counts recover.
* Surgery: Patients with detectable disease undergo resection on week 13. If complete resection is not achieved or if it is deemed impossible, resection must be attempted no later than 3 weeks after consolidation radiotherapy.
* Consolidation: Beginning within 9 days of surgery, patients receive CTX IV over 1 hour on days 1-5 of week 1; VP-16 IV over 1 hour (after CTX infusion) on days 1-5 of week 1 and on days 1-3 of week 4; CBDCA IV over 6 hours on days 1 and 2 of week 4; G-CSF as in induction; and radiotherapy in the absence of disease progression. Patients with complete or partial response after resection and/or radiotherapy proceed to maintenance therapy.
* Maintenance: Patients receive CTX IV over 1 hour on days 1-5 of weeks 0 and 3; VP-16 IV over 1 hour on days 1-5 of weeks 0 and 3 and on days 1-3 of weeks 6 and 9; CBDCA IV over 6 hours on days 1 and 2 of weeks 6 and 9; and G-CSF as in induction. Treatment continues every 12 weeks for 6 courses in the absence of disease progression.

Group D

* Patients receive CBDCA IV over 6 hours on days 1 and 2 and VP-16 IV over 1 hour (after CBDCA infusion) on days 1-3 of weeks 0 and 3. Treatment continues weekly for 6 courses in the absence of disease progression.

Patients are followed every 3 months for 15 months, every 6 months for 1 year, and then annually for 3 years.

PROJECTED ACCRUAL: Not specified

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of Wilms' tumor

  * Eligible subtypes:

    * Favorable histologies
    * Anaplastic histologies
    * Clear cell sarcoma of the kidney
    * Rhabdoid tumor of the kidney
* Relapsed disease after entry on protocol NWTS-5 (NWTS-Q9401)

PATIENT CHARACTERISTICS:

Age:

* 21 and under at original diagnosis

Performance status:

* Not specified

Life expectancy:

* At least 4 weeks

Hematopoietic:

* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times normal
* SGOT or SGPT less than 2.5 times normal

Renal:

* Creatinine no greater than 1.5 times normal OR
* Creatinine clearance or GFR at least 70 mL/min

Cardiovascular:

* Shortening fraction at least 27% by echocardiogram OR
* Ejection fraction greater than 50% by echocardiogram or MUGA scan

Other:

* Not pregnant
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* At least 2 weeks since prior chemotherapy and recovered

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No prior therapy for relapsed Wilms' tumor
* Recovered from the toxic effects of any other prior therapy

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 203 (Actual)
Dates: Start 1996-01; Primary Completion 2002-06 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Event free survival | 2 years
  To determine the two-year second event-free survival percentage for children who relapse following initial therapy with nephrectomy only following treatment with vincristine and dactinomycin, with or without doxorubicin, depending upon the site of relapse and presence or absence of microscopic residual disease.

SECONDARY OUTCOMES:
Event Free Survival | 2 years
  To determine if the two-year second event-free survival percentage for children who relapse following initial treatment with Regimen EE-4A who do not have loss of heterozygosity of markers for chromosome 16q, 1p or increased DNA content in tumor cells is not less than 40% higher than that of similar patients who have loss of heterozygosity for chromosome 16q, 1p or increased DNA content following treatment with intensive chemotherapy using doxorubicin, etoposide, cyclophosphamide and carboplatin, and radiation therapy to sites of microscopic or gross residual disease.
Post-relapse survival | 4 years
  To determine if the four-year post-relapse survival percentage for children who relapse following initial treatment with Regimen DD - 4A who do not have loss of heterozygosity of markers for chromosome 16q, 1p or increased DNA content in tumor cells is not less than 40% higher than that of similar patients who have loss of heterozygosity for chromosome 16q, 1p or increased DNA content following treatment with intensive chemotherapy using etoposide, cyclophosphamide and carboplatin.
Response rate
  To determine if the response rate (CR + PR) of clear cell sarcoma of the kidney and diffuse anaplastic Wilms tumor to the combination of carboplatin and etoposide each exceed 20%.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M. Green, MD, Study Chair — Roswell Park Cancer Institute
Locations (235):
- United States (206):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - University of South Alabama Medical Center, Mobile, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Jonathan Jaques Children's Cancer Center, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital of Oakland, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital at Stanford, Palo Alto, California
  - Sutter Cancer Center, Sacramento, California
  - University of California Davis Medical Center, Sacramento, California
  - Kaiser Permanente Medical Center/Kaiser Foundation Hospital - San Diego, San Diego, California
  - Children's Hospital San Diego, San Diego, California
  - Kaiser Permanente Medical Center - San Francisco Geary Campus, San Francisco, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Children's Hospital of Denver, Denver, Colorado
  - Childhood Hematology/Oncology Associates, Denver, Colorado
  - Presbyterian-St Luke's Medical Center, Denver, Colorado
  - University of Connecticut Health Center, Farmington, Connecticut
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Alfred I. Dupont Institute, Wilmington, Delaware
  - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Shands Hospital and Clinics, University of Florida, Gainesville, Florida
  - Joe DiMaggio Children's Hospital at Memorial, Hollywood, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami-Jackson Memorial Hospital, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Nemours Children's Clinic-Orlando, Orlando, Florida
  - Sacred Heart Children's Hospital, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Tampa Children's Hospital, Tampa, Florida
  - St. Mary's Hospital, West Palm Beach, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Children's Healthcare of Atlanta - Scottish Rite, Atlanta, Georgia
  - Medical College of Georgia Comprehensive Cancer Center, Augusta, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Memorial Health University Medical Center, Inc., Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Mountain States Tumor Institute, Boise, Idaho
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Hope Children's Hospital, Oak Lawn, Illinois
  - Lutheran General Hospital, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - St. Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Raymond Blank Memorial Hospital for Children, Des Moines, Iowa
  - John Stoddard Cancer Center, Des Moines, Iowa
  - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Wesley Medical Center, Wichita, Kansas
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - Ochsner Clinic, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Marlene and Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Floating Hospital for Children, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Massachusetts Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - St. John Hospital and Medical Center, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Spectrum Health and DeVos Children's Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - St. Mary's/Duluth Clinic Cancer Center, Duluth, Minnesota
  - Children's Hospitals and Clinics - Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Children's Hospitals and Clinics of Minnesota, Saint Paul, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - Children's Hospital of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - Atlantic Health System, Summit, New Jersey
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Cancer Center of Albany Medical Center, Albany, New York
  - Brooklyn Hospital Center, Brooklyn, New York
  - State University of New York Health Science Center at Brooklyn College of Medicine, Brooklyn, New York
  - Brookdale University Hospital and Medical Center, Brooklyn, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - North Shore University Hospital, Manhasset, New York
  - Schneider Children's Hospital, New Hyde Park, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Columbia Presbyterian Hospital, New York, New York
  - James P. Wilmot Cancer Center, Rochester, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Albert Einstein Clinical Cancer Center, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Saint Joseph's Health System, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Healthcare, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - East Carolina University School of Medicine, Greenville, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Dakota Cancer Institute, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Children's Hospital of Columbus, Columbus, Ohio
  - Children's Medical Center - Dayton, Dayton, Ohio
  - Toledo Children's Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Forum Health-Tod Childrens Hospital, Youngstown, Ohio
  - Children's Hospital of Oklahoma, Oklahoma City, Oklahoma
  - CCOP - Oklahoma, Tulsa, Oklahoma
  - Natalie Warren Bryant Cancer Center, Tulsa, Oklahoma
  - Doernbecher Children's Hospital, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Palmetto Health South Carolina Cancer Center, Columbia, South Carolina
  - Children's Hospital of Greenville Hospital System, Greenville, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sioux Valley Hospital, Sioux Falls, South Dakota
  - East Tennessee State University Cancer Center at JCMC, Johnson City, Tennessee
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center School of Medicine, Amarillo, Texas
  - Children's Hospital of Austin, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - San Antonio Military Pediatric Cancer and Blood Disorders Center, Lackland Air Force Base, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Methodist Health Care System, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Vermont Cancer Center, Burlington, Vermont
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Naval Medical Center, Portsmouth, Portsmouth, Virginia
  - Massey Cancer Center, Richmond, Virginia
  - Carilion Medical Center for Children, Roanoke, Virginia
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Cooperative, Seattle, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Mary Bridge Children's Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University - Charleston, Charleston, West Virginia
  - Cabell-Huntington Hospital, Inc, Huntington, West Virginia
  - West Virginia University Hospitals, Morgantown, West Virginia
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (6):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Children's Hospital, Brisbane, Queensland
  - Women's and Children's Hospital, North Adelaide, South Australia
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (16):
  - Alberta Children's Hospital, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Children's Health and Rehabilitation Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - Children's Hospital, Hamilton, Ontario
  - Children's Hospital of Western Ontario, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - McGill University Health Center - Montreal Children's Hospital, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Laval University Medical Center, Sainte-Foy, Quebec
  - Centre Hospitalier de L'Universite Laval, Sainte-Foy, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Academisch Ziekenhuis Groningen, Groningen, Netherlands
- Starship Children's Hospital, Auckland, New Zealand
- Puerto Rico (2):
  - University of Puerto Rico School of Medicine Medical Sciences Campus, San Juan
  - San Jorge Childrens Hospital, Santurce
- Switzerland (3):
  - Swiss Pediatric Oncology Group Bern, Bern
  - Swiss Pediatric Oncology Group Geneva, Geneva
  - Swiss Pediatric Oncology Group Lausanne, Lausanne

REFERENCES:
- [Background] Kalapurakal JA, Perlman EJ, Seibel NL, Ritchey M, Dome JS, Grundy PE. Outcomes of patients with revised stage I clear cell sarcoma of kidney treated in National Wilms Tumor Studies 1-5. Int J Radiat Oncol Biol Phys. 2013 Feb 1;85(2):428-31. doi: 10.1016/j.ijrobp.2012.04.023. Epub 2012 Jun 1. PMID 22658515
- [Result] Green DM, Cotton CA, Malogolowkin M, Breslow NE, Perlman E, Miser J, Ritchey ML, Thomas PR, Grundy PE, D'Angio GJ, Beckwith JB, Shamberger RC, Haase GM, Donaldson M, Weetman R, Coppes MJ, Shearer P, Coccia P, Kletzel M, Macklis R, Tomlinson G, Huff V, Newbury R, Weeks D. Treatment of Wilms tumor relapsing after initial treatment with vincristine and actinomycin D: a report from the National Wilms Tumor Study Group. Pediatr Blood Cancer. 2007 May;48(5):493-9. doi: 10.1002/pbc.20822. PMID 16547940
- [Derived] Ehrlich PF, Anderson JR, Ritchey ML, Dome JS, Green DM, Grundy PE, Perlman EJ, Kalapurakal JA, Breslow NE, Shamberger RC. Clinicopathologic findings predictive of relapse in children with stage III favorable-histology Wilms tumor. J Clin Oncol. 2013 Mar 20;31(9):1196-201. doi: 10.1200/JCO.2011.41.1165. Epub 2013 Feb 4. PMID 23382471